CLINICAL TRIAL: NCT01128816
Title: A Multi-Centre, Randomized Study to Assess the Effects of Adaptive Servo Ventilation (ASV) on Survival and Frequency of Hospital Admissions in Patients With Heart Failure (HF) and Sleep Apnea (SA)-The ADVENT-HF Trial
Brief Title: Effect of Adaptive Servo Ventilation (ASV) on Survival and Hospital Admissions in Heart Failure
Acronym: ADVENT-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Philips Global Field Safety Notice for PAP Devices & Ventilators, June 14, 2021 (June 15, 2021 censor date for trial). Patient final visits and collection of endpoints prior to censor date continued to March 31, 2022.
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Philips Respironics (Industry)
Responsible Party: Principal Investigator, Douglas Bradley, Study Chairman, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADVENT-HF trial
Record Dates: First submitted 2010-04-26; First posted 2010-05-24 (Estimated); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Sleep Apnea; Heart Failure
Keywords: obstructive sleep apnea; central sleep apnea; heart failure; congestive heart failure; adaptive servo ventilation; ASV
MeSH Terms: conditions — Sleep Apnea Syndromes; Heart Failure; Sleep Apnea, Obstructive; Sleep Apnea, Central

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard HF therapy (No Intervention): Subjects will receive optimal standard therapy for heart failure conforming to national guidelines as determined by the referring cardiologist
- Standard therapy for HF + ASV (Active Comparator): Subjects will receive treatment with Adaptive Servo Ventilation in addition to optimal standard therapy for heart failure conforming to national guidelines, as determined by the referring cardiologist
  Interventions: Device: Adaptive Servo Ventilation

INTERVENTIONS:
Device: Adaptive Servo Ventilation — BiPAP autoSV ADVANCED device worn nightly during sleep
  Other Names: BiPAP autoSV ADVANCED; ASV; Respironics
  Arms: Standard therapy for HF + ASV

SUMMARY:
Sleep Apnea (SA) is a disorder that causes pauses in breathing during sleep that expose the heart to oxygen deprivation. It is common in patients with heart failure (HF) where it is associated with increased risk of hospitalizations and death. It is not known however whether treating SA reduces these risks. This study is looking at whether a respiratory device known as Adaptive Servo Ventilation (ASV) can reduce the rate of cardiovascular hospitalizations and death in subjects with HF and SA. Study subjects will randomly receive either their regular medications OR their regular medications plus ASV. They will be followed for approximately 5 years and information relevant to their health will be collected and compared.

ELIGIBILITY:
Inclusion Criteria:

* American Heart Association Stage B-D Heart failure due to ischemic, idiopathic or hypertensive causes, present for at least 3 months
* Left Ventricular Ejection Fraction ≤ 45 %
* Optimal medical therapy for heart failure
* No change in active cardiac medications for 2 weeks prior to randomization, beta-blockers must be started 3 months prior to randomization
* Sleep apnea with an AHI ≥ 15. Subjects with obstructive sleep apnea must also have an Epworth Sleepiness Scale score of ≤ 10 and no or mild daytime sleepiness
* Written informed consent

Exclusion Criteria:

* Heart failure due to primary valvular heart disease
* Presence of moderate to severe mitral insufficiency due to intrinsic mitral valve disease
* Hypertrophic obstructive or restrictive or post partum cardiomyopathy
* Exercise capacity limited by class IV angina pectoris
* Acute MI, cardiac surgery, PCI, AICD, or CRT within 3 months of randomization
* Active myocarditis
* Planned AICD or CRT
* Presence of a left-ventricular assist device
* Transplanted heart or expected to receive a transplanted heart within the next 6 months
* Pregnancy
* Current use of ASV or CPAP or mandibular advancement device for treatment of sleep apnea or treated with any investigational therapy during the last 4 weeks (including approved therapies being used in unapproved indications)
* A clinical history that would interfere with the objectives of this study or that would in the investigator's opinion preclude safe conclusion of the study
* Any other medical, social, or geographical factor, which would make it unlikely that the patient will comply with the study procedures (e.g. alcohol abuse, lack of permanent residence, severe depression, disorientation, distant location, or history of non-compliance)
* Any contraindication to ASV therapy as detailed in the device provider manual

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 732 (Actual)
Dates: Start 2010-05; Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
The time to the composite outcome of death or first CV hospital admission or new onset atrial fibrillation/flutter requiring anti-coagulation but not hospitalization or delivery of an appropriate shock from an ICD not resulting in hospitalization. | The expected study follow-up period is five years
  The study will end once 540 primary endpoints have occurred. The maximum follow-up period for all randomized subjects is 5 years.

SECONDARY OUTCOMES:
Time to death from any cause | The expected study follow-up period is 5 years
  The study will end once 540 primary endpoints have occurred.
Number of cardiovascular hospitalizations per year of follow-up | The minimum time of follow-up is expected to be 2 years. The maximum time of follow-up is expected to be 5 years
Number of days alive not hospitalized | Time from randomization to censoring (death, primary event or end of study)
  The number of days the patient is hospitalized are subtracted from the total number of days in the study from randomization. This number will be compared between the 2 groups.
Changes in left ventricular function | 6 months from randomization
  Changes in LV function will be assessed by echocardiography at baseline and at 6 months post randomization
Changes in plasma BNP levels | 6 months from randomization
  Changes in plasma NT-proBNP levels will be assessed at baseline and at 6 months post randomization
Cardiac resynchronization therapy or defibrillator implantations | Average number of days until first cardiac resynchronization or first defibrillator implantation
  The average number of days from randomization to the first occurrence of CRT or defibrillator implantation will be calculated and compared between each treatment arm.
Changes in 6 minute walk test distance | 6 months from randomization
  Changes in the 6-minute walk distance between baseline and 6 months will be compared between the 2 groups
Percentage of patients with changes in stages of heart failure and functional class | Values obtained at study termination will be compared to those obtained at randomization
  New York Heart Association classification and AHA/ACC Stages of Heart Failure will be assessed at each visit.
Changes in apnea/hypopnea index | 1 month from randomization
Changes in Quality of life assessments | Assessments made at baseline, 1, 6, 12 and every 6 months thereafter
  Minnesota living with Heart Failure Questionnaire and Epworth Sleepiness Scale will be used. Scores will be compared between the 2 groups.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Bradley, M.D., Study Chair — Toronto Rehabilitation Institute
Locations (49):
- United States (3):
  - University of Arizona/Southern Arizona VA Health Care System, Tucson, Arizona
  - Glacier View Research Institute, Kalispell Regional Medical Center, Kalispell, Montana
  - MetroHealth Medical Centre, Cleveland, Ohio
- Brazil (4):
  - Pronto Socorro Cardiologico de Pernambuco, Recife, Pernambuco
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo
  - CDEC Brasil - Centro de Desenvolvimento em Estudos Clínicos Brasil, São Paulo, São Paulo
  - Instituto do Coração do Hospital das Clínicas da FMUSP, São Paulo, São Paulo
- Canada (13):
  - Vancouver General Hospital/UBC/VCHA, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Capital District Health Authority, Halifax, Nova Scotia
  - McMaster University Medical Centre, Hamilton Health Sciences, Hamilton, Ontario
  - Kingston General Hospital Sleep Disorders Laboratory/Queen's University, Kingston, Ontario
  - St. Mary's General Hospital, Kitchener, Ontario
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - University of Ottawa-Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network/TRI/Mount Sinai, Toronto, Ontario
  - Hôpital Hôtel-Dieu du CHUM, Montreal, Quebec
  - McGill University Health Centre, Glen Site, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec- Université Laval, Québec, Quebec
- France (7):
  - Centre Hospitalier de Béziers, Béziers
  - Pole d'exploration de L' apnée du sommeil, Nouvelle Clinique Bel Air, Bordeaux
  - Groupe Hospitalier Ambroise Paré, AP-HP, Boulogne-Billancourt
  - Hôpital Antoine Béclère, AP-HP, Clamart
  - Laboratoire d'Explorations Fonctionnelles Cardio-Respiratoires, Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Hôpital Bichat- Claude Bernard, AP-HP, Paris
  - Groupe Hospitalier Pitié-Salpêtrière Charles Foix, AP-HP, Paris
- Germany (2):
  - University of Regensburg, Regensburg, Bavaria
  - Wissenschaftliches Institut Bethanien e.V., Solingen
- Italy (5):
  - ASST Franciacorta, Ospedale di Chiari, Chiari, BS
  - Prima Medicina-Spedali Civili, Brescia
  - Istituto Auxologico Italiano - Ospedale San Luca, Milan
  - Istituto Scientifico di Montescano, Istituti Clinici Scientifici Maugeri (ICS Maugeri), Pavia
  - Istituto Scientifico di Veruno, Istituti Clinici Scientifici Maugeri, Veruno
- Japan (5):
  - Saiseikai Futsukaichi Hospital, Fukuoka
  - Kyoto University Hospital, Kyoto
  - Toranomon Hospital, Tokyo
  - Juntendo University School of Medicine, Tokyo
  - Tokyo Medical University Hospital, Tokyo
- Spain (9):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Arnau de Vilanova, Lleida
  - Fundación Jiménez Diaz-CAPIO, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Rio Hortega, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza
  - Hospital Universitario Txagorritxu, Vitoria-Gasteiz, Álava
- The Sleep Disorders Centre -Nuffield House, Guy's Hospital, London, United Kingdom

REFERENCES:
- [Derived] Horvath CM, Fisser C, Floras JS, Sossalla S, Wang S, Tomlinson G, Rankin F, Yatsu S, Ryan CM, Bradley TD, Arzt M; ADVENT-HF Investigators. Nocturnal Cardiac Arrhythmias in Heart Failure With Obstructive and Central Sleep Apnea. Chest. 2024 Dec;166(6):1546-1556. doi: 10.1016/j.chest.2024.08.003. Epub 2024 Aug 20. PMID 39168180
- [Derived] Bradley TD, Logan AG, Lorenzi Filho G, Kimoff RJ, Duran Cantolla J, Arzt M, Redolfi S, Parati G, Kasai T, Dunlap ME, Delgado D, Yatsu S, Bertolami A, Pedrosa R, Tomlinson G, Marin Trigo JM, Tantucci C, Floras JS; ADVENT-HF Investigators. Adaptive servo-ventilation for sleep-disordered breathing in patients with heart failure with reduced ejection fraction (ADVENT-HF): a multicentre, multinational, parallel-group, open-label, phase 3 randomised controlled trial. Lancet Respir Med. 2024 Feb;12(2):153-166. doi: 10.1016/S2213-2600(23)00374-0. Epub 2023 Dec 21. PMID 38142697
- [Derived] Perger E, Inami T, Lyons OD, Alshaer H, Smith S, Floras JS, Logan AG, Arzt M, Duran Cantolla J, Delgado D, Fitzpatrick M, Fleetham J, Kasai T, Kimoff RJ, Leung RST, Lorenzi Filho G, Mayer P, Mielniczuk L, Morrison DL, Parati G, Parthasarathy S, Redolfi S, Ryan CM, Series F, Tomlinson GA, Woo A, Bradley TD; ADVENT-HF Investigators. Distinct Patterns of Hyperpnea During Cheyne-Stokes Respiration: Implication for Cardiac Function in Patients With Heart Failure. J Clin Sleep Med. 2017 Nov 15;13(11):1235-1241. doi: 10.5664/jcsm.6788. PMID 29065956